CLINICAL TRIAL: NCT00662272
Title: Randomized, Double Blind, Controlled Phase I Trial of the Safety, Tolerability and Immunogenicity of Fluzone® Inactivated Trivalent Influenza Virus Vaccine Administered With Ascending Doses of JVRS-100 Adjuvant
Brief Title: Safety and Efficacy Study of Fluzone® Vaccine Combined With Different Doses of JVRS-100 Adjuvant
Acronym: H-100-001
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Colby Pharmaceutical Company (Industry)
Responsible Party: Maggie Sisti, Juvaris BioTherapeutics, Inc.
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: H-100-001
Record Dates: First submitted 2008-04-15; First posted 2008-04-21 (Estimated); Last update posted 2010-03-17 (Estimated); Status verified 2010-03

CONDITIONS: Influenza
Keywords: Flu; Influenza vaccine; Adjuvant; Safety of an adjuvanted vaccine; Immune response to an adjuvanted vaccine
MeSH Terms: conditions — Influenza, Human | interventions — Adjuvants, Pharmaceutic; Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): Arm includes treatment with Fluzone® vaccine mixed with study product JVRS-100 adjuvant
  Interventions: Biological: Fluzone vaccine with JVRS-100 adjuvant
- 2 (Active Comparator): Arm includes treatment with half adult dose of Fluzone® vaccine
  Interventions: Biological: Fluzone vaccine
- 3 (Active Comparator): Arm includes treatment with full adult dose Fluzone® vaccine
  Interventions: Biological: Fluzone vaccine

INTERVENTIONS:
Biological: Fluzone vaccine with JVRS-100 adjuvant — One vaccination on Day 0 with Fluzone vaccine at 22.5µg mixed with JVRS-100 adjuvant at one of four dose levels (7.5µg, 25µg, 75µg, 225µg) given by IM injection in the upper deltoid.
  Other Names: Fluzone vaccine; adjuvant
  Arms: 1
Biological: Fluzone vaccine — One vaccination on Day 0 with Fluzone vaccine at 22.5µg given by IM injection in the upper deltoid.
  Other Names: Flu vaccine
  Arms: 2
Biological: Fluzone vaccine — One vaccination on Day 0 with Fluzone vaccine at 45µg given by IM injection in the upper deltoid.
  Other Names: Flu vaccination
  Arms: 3

SUMMARY:
This study is designed to assess safety, tolerability and immunogenicity of Fluzone® vaccine with four dose levels of JVRS-100 adjuvant compared to Fluzone® vaccine alone in healthy adults 18-49 years of age.

DETAILED DESCRIPTION:
The purpose of this trial is to evaluate the safety and tolerability of graded, ascending doses of JVRS-100 adjuvant when administered in combination with a vaccine antigen.

ELIGIBILITY:
Inclusion Criteria:

* able to understand the study and provide written informed consent
* be age 18 to 49 years
* be in good general health, without significant medical history, physical examination findings, or abnormal laboratory results
* be available for the study duration, including all planned follow-up visits
* female subjects of child bearing potential must not be pregnant and agree to be correctly using an efficacious hormonal method of contraception or intrauterine device for at least 1 month before the study and during the study

Exclusion Criteria:

* have allergy to eggs or other components of the vaccine
* have had an influenza vaccine within 3 years preceding the screening visit
* have a history of severe reaction of any kind to conventional influenza vaccines
* have or suspected immunodeficiency disorder, including leukemia, lymphoma, generalized malignancy, or treatment with immunosuppressive medications, including corticosteroids, alkylating agents, antimetabolites, or radiation therapy
* have a history of an autoimmune disorder, including systemic lupus, rheumatoid arthritis, scleroderma, other collagen vascular disease, multiple sclerosis, etc. Psoriasis limited to cutaneous manifestations is not an exclusion criterion.
* have prior history of anaphylaxis to foods, hymenoptera stings, vaccines or drugs
* have had transfusion of blood or treatment with any blood product, including intramuscular or intravenous serum globulin within 3 months of the Screening Visit or anticipated through the study period
* have received another vaccine within 30 days preceding the screening visit or anticipated through the study period
* have participation in another clinical trial within 60 days of the screening visit
* have a positive serum or urine pregnancy test prior to vaccination or plan on a pregnancy during study period
* have abnormalities on laboratory assessment
* be seropositive to HIV or HCV or positive for HBsAg
* be positive for anti-nuclear antibodies
* have a physical examination indicating any clinically significant medical condition
* have a body temperature >38.1°C (100.6°F) or acute illness within 3 days prior to vaccination
* intention to travel out of the area prior to the study visit on Day 28 of the study
* have a history of excessive alcohol consumption, drug abuse, significant psychiatric illness
* have the intention to increase normal exercise routine, participate in contact sports or strenuous weight lifting or to initiate vigorous exercise from Screening until after Day 28 of the study

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 128 (Actual)
Dates: Start 2008-06; Primary Completion 2008-10 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Comparison of adverse events between treatment groups | Active Study Duration
Dose-response analysis of HAI geometric mean titers (GMT) | 5 time points

SECONDARY OUTCOMES:
Safety endpoints include between treatment group analyses of all safety parameters as described for the primary endpoint for each ascending dose cohort. | 2 periods
Seroprotection and seroconversion rates to various antigens, distribution of antibody titers, duration of HAI antibody titers, and assessment of cross-reactive HAI responses against "drifted" strains. | 5 time points

CONTACTS AND LOCATIONS:
Overall Officials: Thomas P Monath, MD, Study Director — Medical Monitor for Juvaris
Locations (2):
- United States (2):
  - Miami Research Associates, Miami, Florida
  - Johnson County Clin-Trials, Lenexa, Kansas

REFERENCES:
- [Background] Betts RF, Treanor JJ. Approaches to improved influenza vaccination. Vaccine. 2000 Feb 25;18(16):1690-5. doi: 10.1016/s0264-410x(99)00508-3. PMID 10689150
- [Background] Thompson WW, Shay DK, Weintraub E, Brammer L, Cox N, Anderson LJ, Fukuda K. Mortality associated with influenza and respiratory syncytial virus in the United States. JAMA. 2003 Jan 8;289(2):179-86. doi: 10.1001/jama.289.2.179. PMID 12517228
- [Background] Monto AS, Kioumehr F. The Tecumseh Study of Respiratory Illness. IX. Occurence of influenza in the community, 1966--1971. Am J Epidemiol. 1975 Dec;102(6):553-63. doi: 10.1093/oxfordjournals.aje.a112193. PMID 1202957
- [Background] Barker WH. Excess pneumonia and influenza associated hospitalization during influenza epidemics in the United States, 1970-78. Am J Public Health. 1986 Jul;76(7):761-5. doi: 10.2105/ajph.76.7.761. PMID 3717461
- [Background] Glezen WP. Serious morbidity and mortality associated with influenza epidemics. Epidemiol Rev. 1982;4:25-44. doi: 10.1093/oxfordjournals.epirev.a036250. No abstract available. PMID 6754408
- [Background] Pfleiderer M, Lower J, Kurth R. Cold-attenuated live influenza vaccines, a risk-benefit assessment. Vaccine. 2001 Dec 12;20(5-6):886-94. doi: 10.1016/s0264-410x(01)00386-3. PMID 11738754
- [Background] Hilleman MR. Realities and enigmas of human viral influenza: pathogenesis, epidemiology and control. Vaccine. 2002 Aug 19;20(25-26):3068-87. doi: 10.1016/s0264-410x(02)00254-2. PMID 12163258
- [Background] CBER. Guidance for Industry. Clinical Data Needed to Support the Licensure of Seasonal Inactivated Influenza Vaccines. May 2007. Available at hhtp://www.fda.gov/cber/guidelines.htm
- [Background] Advisory Committee on Immunization Practices; Smith NM, Bresee JS, Shay DK, Uyeki TM, Cox NJ, Strikas RA. Prevention and Control of Influenza: recommendations of the Advisory Committee on Immunization Practices (ACIP). MMWR Recomm Rep. 2006 Jul 28;55(RR-10):1-42. PMID 16874296
- [Background] de Jong JC, Palache AM, Beyer WE, Rimmelzwaan GF, Boon AC, Osterhaus AD. Haemagglutination-inhibiting antibody to influenza virus. Dev Biol (Basel). 2003;115:63-73. PMID 15088777
- [Background] Beyer WE, Palache AM, Luchters G, Nauta J, Osterhaus AD. Seroprotection rate, mean fold increase, seroconversion rate: which parameter adequately expresses seroresponse to influenza vaccination? Virus Res. 2004 Jul;103(1-2):125-32. doi: 10.1016/j.virusres.2004.02.024. PMID 15163500
- [Background] Banzhoff A, Nacci P, Podda A. A new MF59-adjuvanted influenza vaccine enhances the immune response in the elderly with chronic diseases: results from an immunogenicity meta-analysis. Gerontology. 2003 May-Jun;49(3):177-84. doi: 10.1159/000069172. PMID 12679609
- [Background] Amai M, Nojima M, Yuki Y, Kiyono H, Nagamura F. A review of criteria strictness in "Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials". Vaccine. 2023 Aug 31;41(38):5622-5629. doi: 10.1016/j.vaccine.2023.07.072. Epub 2023 Aug 1. PMID 37532612